CLINICAL TRIAL: NCT00419757
Title: A 12-week, Randomised, Double Blind, Active-controlled, Multi-centre, Phase IIIB Study Comparing the Efficacy and Safety of SYMBICORT® pMDI 160/4.5 mg x 2 Actuations Twice Daily Versus Budesonide HFA pMDI 160 mg x 2 Actuations Twice Daily, in Adult/Adolescent (> 12 Yrs) Hispanic Subjects With Asthma
Brief Title: An Efficacy Study Comparing SYMBICORT® Pressurised Metered Dose Inhaler (pMDI) With Budesonide Hydrofluoroalkanes (HFA) pMDI, in Hispanic Subjects With ICS Dependent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5896C00021
Record Dates: First submitted 2007-01-05; First posted 2007-01-09 (Estimated); Results first posted 2012-08-27 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: Asthma
Keywords: Moderate asthma; Severe asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Formoterol Fumarate; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Symbicort (Active Comparator): SYMBICORT® pMDI 160/4.5 μg x 2 actuations twice daily
  Interventions: Drug: Budesonide/formoterol (SYMBICORT) pMDI
- Budesonide (Active Comparator): budesonide HFA pMDI 160 μg x 2 actuations twice daily
  Interventions: Drug: Budesonide HFA pMDI

INTERVENTIONS:
Drug: Budesonide/formoterol (SYMBICORT) pMDI — SYMBICORT® pMDI 160/4.5 μg x 2 actuations twice daily
  Arms: Symbicort
Drug: Budesonide HFA pMDI — Budesonide Hydrofluoroalkane (HFA) pressurised metered dose inhaler (pMDI) 160 μg x 2 actuations twice daily
  Arms: Budesonide

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of SYMBICORT® pMDI (a medication approved by the Food and Drug Administration(FDA)) in the Hispanic population.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, Hispanic (self-reported), > 12 years of age
* Moderate to severe asthma requiring treatment with an inhaled corticosteroid
* Diagnosis of asthma for at least 6 months

Exclusion Criteria:

* Subjects requiring treatment with systemic corticosteroids (e.g., oral, parenteral, ocular)
* Any significant disease or disorder that may jeopardize a subject's safety

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christer Hultquist, MD, Study Director — AstraZeneca
Locations (39):
- United States (32):
  - Research Site, Anaheim, California
  - Research Site, Chula Vista, California
  - Research Site, Fresno, California
  - Research Site, Fullerton, California
  - Research Site, Los Angeles, California
  - Research Site, National City, California
  - Research Site, Rancho Cordova, California
  - Research Site, Rancho Mirage, California
  - Research Site, Riverside, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Stockton, California
  - Research Site, Torrance, California
  - Research Site, Pueblo, Colorado
  - Research Site, Largo, Florida
  - Research Site, Miami, Florida
  - Research Site, Naranja, Florida
  - Research Site, North Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Panama City, Florida
  - Research Site, South Miami, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Newburgh, New York
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Boerne, Texas
  - Research Site, El Paso, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Spring, Texas
- Puerto Rico (7):
  - Research Site, Aguas Buenas
  - Research Site, Caquas
  - Research Site, Cidra
  - Research Site, Levittown
  - Research Site, Ponce
  - Research Site, SanJuan
  - Research Site, Trujillo Alto

REFERENCES:
- [Derived] Murphy KR, Uryniak T, Martin UJ, Zangrilli J. The effect of budesonide/formoterol pressurized metered-dose inhaler on predefined criteria for worsening asthma in four different patient populations with asthma. Drugs R D. 2012 Mar 1;12(1):9-14. doi: 10.2165/11630600-000000000-00000. PMID 22329608
- [Derived] Zangrilli J, Mansfield LE, Uryniak T, O'Brien CD. Efficacy of budesonide/formoterol pressurized metered-dose inhaler versus budesonide pressurized metered-dose inhaler alone in Hispanic adults and adolescents with asthma: a randomized, controlled trial. Ann Allergy Asthma Immunol. 2011 Sep;107(3):258-65.e2. doi: 10.1016/j.anai.2011.05.024. Epub 2011 Jul 14. PMID 21875546
- See also: Related Info — http://www.asthmaclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 39 centres in United States enrolled 558 patients with asthma into this study. 308 patients were excluded: 279 for incorrect enrollment/eligibility criteria not fulfilled, 14 for voluntary discontinuations, 2 for development of study specific discontinuation criteria, 2 for adverse events, 10 were lost to follow-up
Pre-assignment Details: Male or female, Hispanic (self-reported), ≥12 years
Groups:
- Symbicort: SYMBICORT® pMDI 160/4.5 μg x 2actuations twice daily
- Budesonide: Budesonide Hydrofluoroalkane (HFA) pressurised metered dose inhaler (pMDI) 160 μg x 2 actuations twice daily
Period: Overall Study
Arm/Group | Symbicort | Budesonide
Started | 127 (Randomized patients) | 123 (Randomized patients)
Completed | 109 (Randomized patients) | 102 (Randomized patients)
Not Completed | 18 | 21
Not completed — Adverse Event | 1 | 4
Not completed — Lost to Follow-up | 1 | 4
Not completed — Withdrawal by Subject | 7 | 1
Not completed — Protocol Violation | 2 | 3
Not completed — Study specific discontinuation criteria | 4 | 8
Not completed — Multiple reasons | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symbicort | Budesonide | Total
Number analyzed (Participants) | 127 | 123 | 250
Age Continuous [Mean (Standard Deviation); unit: Years] | 16.6 (39.8) | 14.9 (37.0) | 15.6 (38.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 80 | 164
  Male | 43 | 43 | 86

OUTCOME MEASURES:

1. Primary Outcome: Morning Peak Expiratory Flow (AM PEF)
Description: Change from baseline (average of daily records over the 14 days of run-in) to the average of daily records over the treatment period of 12 weeks, with baseline value as covariate.
Time Frame: Baseline (run-in) and throughout 12 weeks
Population: Includes all subjects who were randomised, took at least one dose of study medication and contributed sufficient data for the endpoint to be calculated.
Measure: Least Squares Mean (Standard Error); unit: Liters/minutes
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 124 | 119
Liters/minutes | 25.40 (6.0) [lower limit +/-6.0] | 19.90 (6.5) [lower limit +/-6.5]

2. Secondary Outcome: Percentage of Participants With Pre-defined Asthma Events
Description: Asthma Events, defined as any of: decrease in lung function (FEV1 or AM PEF), use of rescue medication over maximum allowed per day, night awakening requiring use of rescue medication, exacerbation of asthma requiring medical assistance, use of not allowed asthma medication
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 127 | 123
Percentage of Participants | 25.20 | 31.70

3. Secondary Outcome: Percentage of Participants With "Withdrawals Due to Pre-defined Asthma Events"
Description: Percentage of participants with "Withdrawals Due to Pre-defined Asthma Events" as recorded in CRF. Includes all subjects who were randomised, took at least one dose of study medication and contributed sufficient data for the endpoint to be calculated.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 96 | 92
Percentage of Participants | 2.10 | 6.50

4. Secondary Outcome: Changes Pre-dose Forced Expiratory Volume in 1 Second (FEV1)
Description: Changes in pre-dose FEV1 from baseline to the average value over the treatment period, with baseline value as covariate. Includes all subjects who were randomised, took at least one dose of study medication and contributed sufficient data for the endpoint to be calculated.
Time Frame: Baseline, 2, 6 and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 124 | 122
Liters | 0.16 (0.03) [lower limit +/-0.03] | 0.11 (0.03) [lower limit +/-0.03]

5. Secondary Outcome: Change From Baseline in a Evening Peak Expiratory Flow (PM PEF)
Description: Change from baseline (average of daily records over the 14 days of run-in) to the average of daily records over the treatment period of 12 weeks with baseline as covariate. Includes all subjects who were randomised, took at least one dose of study medication and contributed sufficient data for the endpoint to be calculated.
Time Frame: Baseline (run-in) and throughout 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/minutes
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 124 | 119
Liters/minutes | 20.60 (6.2) [lower limit +/-6.2] | 15.80 (6.7) [lower limit +/-6.7]

6. Secondary Outcome: Change in Nighttime Asthma Symptom Score From Baseline Through 12 Weeks
Description: Change from baseline in average of daily scores for nighttime asthma over 12 weeks of treatment, with baseline value as covariate.
  Daily scale:
  * 0 = No symptoms
  * 1 = Mild symptoms
  * 2 = Moderate symptoms
  * 3 = Severe symptoms
Time Frame: Baseline (run-in) and throughout 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 125 | 119
Units on a scale | -0.40 (0.01) [lower limit +/-0.01] | -0.30 (0.01) [lower limit +/-0.01]

7. Secondary Outcome: Change in Daytime Asthma Symptom Score From Baseline Through 12 Weeks
Description: Change from baseline in average of daily scores for daytime asthma over 12 weeks of treatment, with baseline value as covariate.
  Daily scale:
  * 0 = No symptoms
  * 1 = Mild symptoms
  * 2 = Moderate symptoms
  * 3 = Severe symptoms
Time Frame: Baseline (run-in) and throughout 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 125 | 119
Units on a scale | -0.40 (0.01) [lower limit +/-0.01] | -0.30 (0.01) [lower limit +/-0.01]

8. Secondary Outcome: Change in Asthma Related Awakenings Free Nights, From Baseline Through 12 Weeks
Description: Change from baseline in percentage of nights with awakenings due to asthma over 12 weeks of treatment, with baseline value as covariate.
Time Frame: Baseline (run-in) and throughout 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of nights
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 125 | 119
Percentage of nights | 5.40 (1.7) [lower limit +/-1.7] | 5.50 (1.9) [lower limit +/-1.9]

9. Secondary Outcome: Change From Baseline in Rescue Medication Use Over 12 Weeks of Treatment
Description: Change from baseline in rescue medication use over 12 weeks of treatment with baseline value as covariate. Includes all subjects who were randomised, took at least one dose of study medication and contributed sufficient data for the endpoint to be calculated.
Time Frame: Baseline (run-in) and throughout 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: puffs/day
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 125 | 119
puffs/day | -0.80 (0.20) [lower limit +/-0.20] | -0.60 (0.20) [lower limit +/-0.20]

10. Secondary Outcome: Change From Baseline in Rescue-free Days Over 12 Weeks of Treatment
Description: Change from baseline in percentage of rescue-free days over 12 weeks of treatment, with baseline value as covariate. Includes all subjects who were randomised, took at least one dose of study medication and contributed sufficient data for the endpoint to be calculated.
Time Frame: Baseline (run-in) and throughout 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 125 | 119
Percentage of days | 19.70 (3.30) [lower limit +/-3.30] | 17.70 (3.50) [lower limit +/-3.50]

11. Secondary Outcome: Change From Baseline in Symptom-free Days Over 12 Weeks of Treatment
Description: Change from baseline in percentage of symptom-free days over 12 weeks of treatment, with baseline value as covariate. Includes all subjects who were randomised, took at least one dose of study medication and contributed sufficient data for the endpoint to be calculated.
Time Frame: Baseline (run-in) and throughout 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 125 | 119
Percentage of days | 24.40 (3.30) [lower limit +/-3.30] | 21.00 (3.50) [lower limit +/-3.50]

12. Secondary Outcome: Subject Global Assessment
Description: The assessment was made using a 5-point Likert scale with 1=much better, 2=somewhat better, 3=comparable, 4=somewhat worse, and 5=much worse transformed to a binary variable with points 1 and 2 combined as "Yes" and points 3, 4, 5 as "No". Percent of Participants that gave positive responses.
Time Frame: Baseline and week 12
Population: as for outcome 1
Measure: Number; unit: Percent of Participants
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 125 | 119
Percent of Participants | 88.70 | 86.30

13. Secondary Outcome: Physician Global Assessment
Description: The assessment was made using a 5-point scale with 1=much better, 2=somewhat better, 3=comparable, 4=somewhat worse, and 5=much worse transformed to a binary variable with points 1and 2 combined as "Yes" and points 3, 4, 5 as "No". Percent of Participants that gave positive responses.
Time Frame: Baseline and week 12
Population: as for outcome 1
Measure: Number; unit: Perscentage of Participants
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 125 | 119
Perscentage of Participants | 92.00 | 84.60

14. Secondary Outcome: Patient Satisfaction With Asthma Medication (PSAM) in Term of Domain: Control Relief Index
Description: Mean scores (6-points scale, where 1-means the most positive opinion and 6-the most negative opinion) were calculated for items in domain. 6-point response options were scored on a 0±100 scale, where 100 represented the highest level of satisfaction and 0 the lowest level of satisfaction.
Time Frame: Week 12
Population: Only subjects 18 years and older, who were randomised, took at least one dose of study medication and contributed sufficient data for the endpoint to be calculated.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 104 | 100
Units on a scale | 87.20 (1.97) [lower limit +/-1.97] | 82.50 (2.08) [lower limit +/-2.08]

15. Secondary Outcome: Patient Satisfaction With Asthma Medication (PSAM) in Term of Domain: Overall Perception of Medication
Description: Mean scores (6 or 5-points scale, where 1-means the most positive opinion and 5/6-the most negative opinion) were calculated for items in domain. 6-point response options were scored on a 0±100 scale, where 100 represented the highest level of satisfaction and 0 the lowest level of satisfaction.
Time Frame: Week 12
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 104 | 100
Units on a scale | 90.67 (1.79) | 86.66 (1.89)

16. Secondary Outcome: Patient Satisfaction With Asthma Medication (PSAM) in Term of Domain: Comparison With Other Medications
Description: Mean scores (5-points scale, where 1-means the most positive opinion and 5-the most negative opinion) were calculated for items in domain. 6-point response options were scored on a 0±100 scale, where 100 represented the highest level of satisfaction and 0 the lowest level of satisfaction.
Time Frame: Week 12
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 104 | 100
Units on a scale | 88.45 (2.34) | 80.60 (2.47)

ADVERSE EVENTS:
Arm/Group | Symbicort | Budesonide
Serious Adverse Events (participants affected / at risk) | 4/127 | 0/123
Other Adverse Events (participants affected / at risk) | 69/127 | 48/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort (N=127) | Budesonide (N=123)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Status Asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort (N=127) | Budesonide (N=123)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Bronchitis (Infections and infestations) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 0
Ear Pain (Ear and labyrinth disorders) | 3 | 0
Headache (Nervous system disorders) | 19 | 14
Influenza (Infections and infestations) | 3 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Nasopharyngitis (Infections and infestations) | 7 | 0
Pain (General disorders) | 3 | 0
Pharyngitis Streptococcal (Infections and infestations) | 3 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pyrexia (General disorders) | 3 | 0
Sinusitis (Infections and infestations) | 0 | 3
Toothache (Gastrointestinal disorders) | 0 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 4
Viral Upper Respiratory Tract Infection (Infections and infestations) | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No